CLINICAL TRIAL: NCT01764464
Title: Gralise® for Spine Surgery Pain (GRASSP): A Partially Enriched, Placebo Controlled, Randomized, Double Blind, Cross-Over Trial of Gralise® for the Treatment of Post Laminectomy Pain Syndrome
Brief Title: GRASSP: Gralise® for Spine Surgery Pain
Acronym: GRASSP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, John Markman, Director, Translational Pain Research, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: RSRB00041904
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Post-laminectomy Pain Syndrome
Keywords: post laminectomy pain syndrome, failed back surgery syndrome
MeSH Terms: conditions — Failed Back Surgery Syndrome | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): 14 day titration (days 1-7 at 600 mg daily Gralise®; days 8-14 at 1200 mg daily Gralise®). 28 day maintenance (1800 mg daily Gralise®). 7 day taper (days 1-4 at 1200 mg daily Gralise®; days 5-7 at 600 mg daily Gralise®). 10 day washout (no intervention). 14 day titration (days 1-7 at 600 mg daily placebo; days 8-14 at 1200 mg daily placebo). 28 day maintenance (1800 mg daily placebo). 7 day taper (days 1-4 at 1200 mg daily placebo; days 5-7 at 600 mg daily placebo).
  Interventions: Drug: Gralise®; Drug: Placebo
- Group B (Other): 14 day titration (days 1-7 at 600 mg daily placebo; days 8-14 at 1200 mg daily placebo). 28 day maintenance (1800 mg daily placebo). 7 day taper (days 1-4 at 1200 mg daily placebo; days 5-7 at 600 mg daily placebo). 10 day washout (no intervention). 14 day titration (days 1-7 at 600 mg daily Gralise®; days 8-14 at 1200 mg daily Gralise®). 28 day maintenance (1800 mg daily Gralise®). 7 day taper (days 1-4 at 1200 mg daily Gralise®; days 5-7 at 600 mg daily Gralise®).
  Interventions: Drug: Gralise®; Drug: Placebo

INTERVENTIONS:
Drug: Gralise® — 14 day titration (days 1-7 at 600 mg daily Gralise®; days 8-14 at 1200 mg daily Gralise®). 28 day maintenance (1800 mg daily Gralise®). 7 day taper (days 1-4 at 1200 mg daily Gralise®; days 5-7 at 600 mg daily Gralise®).
  Other Names: Gralise: Gabapentin ER
Drug: Placebo — 14 day titration (days 1-7 at 600 mg daily placebo; days 8-14 at 1200 mg daily placebo). 28 day maintenance (1800 mg daily placebo). 7 day taper (days 1-4 at 1200 mg daily placebo; days 5-7 at 600 mg daily placebo).
  Other Names: Placebo: inactive pill manufactured to mimic gralise.

SUMMARY:
Evaluate the analgesic benefit of Gralise® for post-laminectomy pain syndrome (PLPS)

ELIGIBILITY:
Inclusion Criteria.

1. Male and female subjects age 18 to 80 years.
2. Primary diagnosis of post-laminectomy pain syndrome (PLPS), defined as having their most severe pain related to a prior history of lumbar surgery including decompressive (e.g. laminectomy) or fusion (e.g. posterior lumbar interbody fusion) procedures performed from the L1-S1 level at least 6 months prior to enrollment.
3. Pain Detect score ≥12, denoting neuropathic pain is probable.
4. At least 50% of present pain intensity is attributed to the lower extremity (Quebec Task Force Grade 3 or 4) on most days.
5. All subjects must be decisionally capable and must give their own consent to be enrolled.

Exclusion Criteria.

1. Lumbar surgery <6 months prior to enrollment
2. Subjects with PLPS and pain free interval (defined as chronic low back pain and radicular symptoms <=3/10) related the indication for their PLPS defining event and a new, acute or subacute symptom pattern (e.g. new disc herniation at an adjacent level as documented by imaging).
3. Subjects regularly taking gabapentin or pregabalin for their chronic pain after spine surgery who do not endorse relief (defined as either minimally, much or very much improved on a 7 point likert scale when asked about these medications' effects).
4. Having another type of pain that is as or more severe than pain associated with PLPS.
5. An average daily pain score of 10 on the NRS scale during either the screening or initial washout period.
6. Concurrent medication that includes antiepileptic drugs (AEDs) (exceptions: pregabalin or gabapentin).
7. Subjects taking concomitant neuropathic pain medication (stable dose for at least 4 weeks) may reduce the number and/or dose of their current pain medications: If the number and/or dose exceed the limits of allowed neuropathic pain medications (refer to Use of Allowed Pain Medication), then the number and/or dose must be reduced to fall within acceptable limits. Concomitant neuropathic pain medication needs to be kept stable during the study.
8. Subjects who have previously not responded to treatment with gabapentin at doses of ≥900 mg/day or pregabalin at doses ≥300 mg/day.
9. Known hypersensitivity to Gralise, or gabapentin, or its ingredients.
10. Dose limiting adverse events to gabapentin; subjects who previously experienced dose-limiting adverse effects that prevented titration of gabapentin to an effective dose.
11. History of alcohol and/or drug abuse in the investigator's judgment, based on subject history and physical examination.
12. Subject who consumes excessive amounts of alcohol, defined as greater than 3 glasses of alcoholic beverages (1 glass is approximately equivalent to: beer [10 ounces], wine [4 ounces], or distilled spirits [1 ounce]) per day on a regular basis.
13. Participation in a clinical trial of an investigational drug or device within 30 days of the screening visit.
14. Gastric reduction surgery.
15. Acute gastrointestinal symptoms such as diarrhea, dyspepsia, or gastric or duodenal ulcers.
16. Malignancy within past 2 years other than basal cell carcinoma.
17. Women who are pregnant or breastfeeding.
18. History of seizure or is at risk of seizure due to head trauma.
19. History of significant cardiovascular, respiratory, endocrine, liver or kidney disease (subjects with renal impairment or creatine clearance <30 ml/min).
20. Any significant medical condition, laboratory abnormality, or psychiatric illness (e.g. depression, mood problems, suicidal thoughts) that would prevent the subject from participating in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Markman, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 53 subjects signed consent and were enrolled in the study. 22 subjects were ineligible after enrollment for the following: did not meet inclusion/exclusion criteria (n=12), withdrew consent during screening period (n=5), non-responder to gabapentinoid during washout period (n=5). A total of 32 subjects were randomized, 25 completed.
Groups:
- Group A (Gralise Then Placebo): 14 day titration (days 1-7 at 600 mg daily Gralise®; days 8-14 at 1200 mg daily Gralise®). 28 day maintenance (1800 mg daily Gralise®). 7 day taper (days 1-4 at 1200 mg daily Gralise®; days 5-7 at 600 mg daily Gralise®). 10 day washout (no intervention). 14 day titration (days 1-7 at 600 mg daily placebo; days 8-14 at 1200 mg daily placebo). 28 day maintenance (1800 mg daily placebo). 7 day taper (days 1-4 at 1200 mg daily placebo; days 5-7 at 600 mg daily placebo).
- Group B (Placebo Then Gralise): 14 day titration (days 1-7 at 600 mg daily placebo; days 8-14 at 1200 mg daily placebo). 28 day maintenance (1800 mg daily placebo). 7 day taper (days 1-4 at 1200 mg daily placebo; days 5-7 at 600 mg daily placebo). 10 day washout (no intervention). 14 day titration (days 1-7 at 600 mg daily Gralise®; days 8-14 at 1200 mg daily Gralise®). 28 day maintenance (1800 mg daily Gralise®). 7 day taper (days 1-4 at 1200 mg daily Gralise®; days 5-7 at 600 mg daily Gralise®).
Period: First Intervention
Arm/Group | Group A (Gralise Then Placebo) | Group B (Placebo Then Gralise)
Started | 16 (Started Gralise) | 16 (Started Placebo)
Completed | 14 (Completed Gralise) | 13 (Completed Placebo)
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Adverse Event | 0 | 2
Not completed — did not receive study drug | 0 | 1
Period: Second Intervention (Cross-over)
Arm/Group | Group A (Gralise Then Placebo) | Group B (Placebo Then Gralise)
Started | 14 (Started Placebo) | 13 (Started Gralise)
Completed | 12 (Completed Placebo) | 13 (Completed Gralise)
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 10 | 23
  >=65 years | 3 | 6 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 9 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 16 | 14 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Numeric Rating Scale (NRS)
Description: Using the Numeric Rating Scale (NRS) (0=no pain, 10=worst pain imaginable).
Time Frame: baseline to 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Gralise: Gralise
- Placebo: Placebo
Arm/Group | Gralise | Placebo
Number analyzed (Participants) | 32 | 32
units on a scale | -0.56 [-2.06 to 0.95] | -0.54 [-2.06 to 0.96]

2. Secondary Outcome: Mean Change in Visual Analog Scale (VAS)
Description: The VAS asks subjects to place a mark indicative of their low back pain during the past day on a 100mm line, with 0mm representing no pain and 100mm representing extreme pain.
Time Frame: baseline to 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Gralise | Placebo
Number analyzed (Participants) | 32 | 32
mm | -0.47 [-2.21 to 1.26] | 0.31 [-1.42 to 2.05]

3. Secondary Outcome: Mean Change in Patient Global Assessment (PGA)
Description: Subjects will be asked to rate their low back pain according to the PGA. PGA is the impact of disease activity. PGA is measured on a 5-point scale, where 1=very good, 2=good, 3=fair, 4=poor, and 5=very poor.
Time Frame: baseline to 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Gralise | Placebo
Number analyzed (Participants) | 32 | 32
units on a scale | -0.04 [-0.11 to 0.04] | -0.00 [-0.08 to 0.07]

4. Secondary Outcome: Mean McGill Pain Questionnaire-2 (MPQ-2)
Description: The McGill Pain questionnaire is 22 questions where patient rate their pain symptoms with each question scaled 0-10 for a total 220 points where a higher score indicates worse outcome.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gralise | Placebo
Number analyzed (Participants) | 27 | 25
units on a scale | 2.97 (1.79) | 3.13 (1.85)

5. Secondary Outcome: Mean Change in Modified Brief Pain Inventory- Short Form (mBPI-sf)
Description: The mBPI is a series of questions that rates the severity and impact of pain on daily function. The questionnaire is made up of 4 pain severity items using the NRS scale, and seven 11-point pain interference scales (0 indicating no interference and 10 indicating complete interference). The scale ranges from 0 to 70. Higher scores indicate worse outcome.
Time Frame: baseline to 6 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Gralise | Placebo
Number analyzed (Participants) | 32 | 32
units on a scale | -0.07 [-0.21 to 0.06] | -0.07 [-0.21 to 0.07]

6. Secondary Outcome: Insomnia Severity Index (ISI)
Description: The ISI has 7 questions with each question ranging from 0-4 for a total of 28 points with higher scores indicating more severe insomnia.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gralise | Placebo
Number analyzed (Participants) | 27 | 25
units on a scale | 16.81 (6.88) | 18.40 (7.34)

ADVERSE EVENTS:
Time Frame: 143 days
Arm/Group | Gralise | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 16/32 | 14/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gralise (N=32) | Placebo (N=32)
Weight gain (General disorders) | 2 | 0
peripheral edema (General disorders) | 2 | 0
Decreased sex drive (General disorders) | 2 | 0
Head cold (General disorders) | 2 | 2
Diaphoretic (General disorders) | 1 | 2
Depression (Psychiatric disorders) | 2 | 1
Anxiety (Psychiatric disorders) | 2 | 2
Euphoria (Psychiatric disorders) | 2 | 0
Increased Pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Muscle Cramps (Musculoskeletal and connective tissue disorders) | 2 | 3
Dizziness (Nervous system disorders) | 4 | 2
Somnolence (Nervous system disorders) | 7 | 0
Headache (Nervous system disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes